CLINICAL TRIAL: NCT04002440
Title: Directed Use of REmote Patient Management System AMia to Achieve Prescribed Dry Weight
Acronym: DREAM-APD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Scripps Health (Other); Home Dialysis Therapies of San Diego (Unknown)
Responsible Party: Principal Investigator, Joachim H. Ix, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 180492
Record Dates: First submitted 2018-10-11; First posted 2019-06-28 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Efficacy; Safety Issues
Keywords: Estimated Dry Weight; Peritoneal Dialysis; AMIA; Sharesource; CCPD; Peritoneal Dialysis Cycler; HomeChoice PRO

STUDY DESIGN:
Intervention Model Description: Participants will be consented and then randomized to one of 2 modality groups; AMIA or HomeChoice PRO. Participants will receive PD care with randomized modality for 6 months, then cross-over to other modality for next 6 months. Nephrologists will see patients once a month. Each visit, the nephrologist will define the patient's desired dry weight (DW) at the subsequent visit. The primary end-point will be the average difference between actual DW vs. prescribed DW. The investigators envision a learning curve with each cycler change, and therefore have set the primary endpoint to average the final 3 visits, rather than using all 6 visits. All solutions and supplies will be from Baxter. Labs will be obtained monthly and quarterly per routine. Dialysis RN will review patients on AMIA twice a week and contact those off target DW and offer interventions to achieve prescribed DW. HomeChoice PRO will record data on a chip analyzed at the end of 6 months to evaluate compliance.
Masking Description: The study is not blinded, as the intervention does not provide an opportunity to blind either the physician or the patient. The PI will be masked to randomization and not involved in patient care or data collection. Statistical analyses will be conducted by Dr. Ronit Katz who is not an investigator for this trial and PI Dr.Joachim Ix after being provided secure study results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AMIA with SHARESOURCE (Active Comparator): For this arm, dialysis nurses will review those patients using the AMIA with SHARESOURCE connectivity platform twice a week and will contact patients who meet certain triggers. They will then offer patients interventions, ie. a change in the preset AMIA ultrafiltration program, in order to achieve prescribed dry weight.
  Interventions: Combination Product: AMIA with SHARESOURCE Connectivity Platform
- HomeChoice PRO (Placebo Comparator): For this arm, routine standard of care for peritoneal dialysis patients will continue using the HomeChoice PRO device. Data regarding treatments will be captured on a chip to be analyzed at the end of 6 months to evaluate compliance with treatments.
  Interventions: Device: HomeChoice PRO

INTERVENTIONS:
Combination Product: AMIA with SHARESOURCE Connectivity Platform — The investigators will conduct a randomized, cross-over study in peritoneal dialysis patients in which patients are randomized to either Home Choice Pro (which remains the most widely used Baxter cycler) versus treatment with the Baxter AMIA automated peritoneal dialysis system with SHARESOURCE connectivity.
  Other Names: Baxter AMIA; SHARESOURCE
  Arms: AMIA with SHARESOURCE
Device: HomeChoice PRO — Usual care
  Other Names: Baxter HomeChoice PRO
  Arms: HomeChoice PRO

SUMMARY:
Among ambulatory peritoneal dialysis patients, does use of the Baxter AMIA peritoneal dialysis cycler with SHARESOURCE connectivity platform achieve dry weight targets better than use of the Baxter Home Choice Pro cycler.

DETAILED DESCRIPTION:
The remote patient management system Baxter AMIA automated peritoneal dialysis system with SHARESOURCE connectivity platform incorporates innovative technology (two-way remote connectivity, touch screen controls, voice guidance) to record patient treatments which are then able to be transmitted to their dialysis clinic for review and monitoring in near real-time. This has tremendous potential clinical utility given the struggles to achieve dry weights for most peritoneal dialysis patients using other systems, where typically, management regarding fluid balance is reviewed and revised only monthly. The new technology is the only device cleared in the US with patient-centric features. Abstracts available have demonstrated that AMIA can improve efficiency of patient training and focus PD nursing time towards proactive tasks to help patients. There has also been insight into how remote patient management systems like AMIA can be used to objectively monitor patient compliance or catheter function above and beyond subjective endorsement from patients. However, with new technology comes new training for patient and staff (nurses, physicians) without understanding if interfacing with this new patient-centric featured technology improves patient-centric clinical outcomes. The new AMIA and SHARESOURCE programs may also require additional nurse and physician provider time to monitor data in real-time and to react to these data, which may incur additional expense to medical practices. Thus, it is imperative to demonstrate the utility of the AMIA and SHARESOURCE programs for important improvement in patient management, which may ultimately translate into improved clinical outcomes (e.g. fewer hospital admissions, less heart failure, improved quality, and length of life).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > 21 years with ESRD on peritoneal dialysis

Exclusion Criteria:

* Unable to commit to 12 months of monitoring.
* Unable to stand safely on scale for weight
* Hospitalization for heart failure, volume overload, or cardiovascular disease within the last 3 months.
* Peritonitis within the past 3 months.
* Not responsible for self-care of peritoneal dialysis (proxy care will be excluded).
* Patients residing in a nursing home or other institutionalized individuals.
* Inability or unwillingness to provide informed consent (lacks decision making capacity)
* Alcohol, substance use, or other social conditions which preclude close follow-up and reliable participation, in the opinion of the primary nephrology physician or study investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
3 month average of difference between the actual vs. prescribed dry weight | 3 months
  The investigators will evaluate the average difference between the actual dry weight vs. prescribed dry weight achieved through use of Baxter AMIA automated peritoneal dialysis system with SHARESOURCE connectivity compared to use of HomeChoicePRO.

SECONDARY OUTCOMES:
Nursing burden related to use of AMIA with SHARESOURCE | 12 months
  The investigators will observe the number of nursing time hours per month dedicated to patient care for patients using AMIA with SHARESOURCE compared to patients using HomeChoicePRO.
Patient Quality of Life while using AMIA with SHARESOURCE: Kidney Disease and Quality of Life -36 questionaire | 12 months
  The investigators will assess quality of life scores using the Kidney Disease and Quality of Life -36 questionaire survey of patients using AMIA with SHARESOURCE compared to patients using HomeChoicePRO. The survey assesses 5 areas pertaining to quality of life on dialysis which include 1) physical component score 2) mental component score 3) burden 4) symptoms 5) effects. Patient answers are compared to their national demographic and reported on a scale of 0-100. The higher the score the better. The scores for each component will be reported and tracked separately.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim H Ix, MD, MAS, Principal Investigator — University of California, San Diego; Bethany E Karl, DO, Study Director — University of California, San Diego
Locations (2):
- United States (2):
  - Home Dialysis Therapies of San Diego, Chula Vista, California
  - Home Dialysis Therapies of San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: Undecided